CLINICAL TRIAL: NCT03351413
Title: SAFE-LiFE to Prevent Falls Among Older Fallers
Brief Title: Preventing Falls Among Older Fallers to Test the Effect of LIVE-LiFE, a Home-Based, Tailored Fall Prevention Program
Acronym: LIVE-LiFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00141297
Record Dates: First submitted 2017-11-20; First posted 2017-11-22 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Fall Prevention
Keywords: Fall Prevention; Older Adults

STUDY DESIGN:
Intervention Model Description: Single-blind, two group randomized pilot trial. Randomization is 2:1 (27 intervention, 13 control). Participants have a chance of being in the LIVE-LiFE group or the control group.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): LIVE-LiFE to Prevent Falls Among Older Fallers Intervention, which is an individually tailored program at the participant's home spaced across 12 weeks including:
  * Home safety assessment and risk reduction strategies; incorporating strength and balance training into daily habits vision screening and referral; and education about fear of falling and falls
  * Home repairs, modifications, and low cost assistive devices to address unsafe home environments increasing fall risk
  * Medication review and feedback concerning medications with increased fall risk
  Interventions: Other: LIVE-LiFE to Prevent Falls Among Older Fallers
- Control (No Intervention): - An individualized fall risk assessment provided to participant and their primary care provider

INTERVENTIONS:
Other: LIVE-LiFE to Prevent Falls Among Older Fallers — LIVE-LiFE Intervention: Individually tailored program at the participant's home spaced across 12 weeks including:
  * Home safety assessment and risk reduction strategies; incorporating strength and balance training into daily habits vision screening and referral; and education about fear of falling and falls
  * Home repairs, modifications, and low cost assistive devices to address unsafe home environments increasing fall risk
  * Medication review and feedback concerning medications with increased fall risk
  Measurement intervals: Baseline, 4 months, 8 months (with $25 gift card given at each visit for your time)
  Other Names: LIVE-LiFE
  Arms: Intervention

SUMMARY:
Purpose: To test the effect of LIVE-LiFE, a home-based, tailored fall prevention program for older adults with a high risk for falling.

Study Type: Single-blind, two group randomized pilot trial. Randomization is 2:1 (27 intervention, 13 control). Participants have a chance of being in the LIVE-LiFE group or the control group.

Safe-LiFE Group: Individually tailored intervention at the participant's home spaced across 12 weeks including:

* Home safety assessment and risk reduction strategies; incorporating strength and balance training into daily habits vision screening and referral; and education about fear of falling and falls
* Home repairs, modifications, and low cost assistive devices to address unsafe home environments increasing fall risk
* Medication review and feedback concerning medications with increased fall risk

Control Group:

• An individualized fall risk assessment provided to participant and their primary care provider

Sample: 40 community-dwelling older adults in Baltimore City or County

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 70 or older
* Self-report of 2 or more falls in the past 12 months OR 1 fall causing injury in the past 12 months

Exclusion Criteria:

* Moderate-severe memory problems
* No conversational English
* Not able to stand
* Resident in a nursing home or assisted living facility
* Hospitalized > 3 times in the last year
* Terminally ill (<1 year expected survival)
* Receiving active cancer treatment

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Times Up and Go Test | Baseline to 16 weeks
  A test used to assess the length of time it takes a person to get out of a chair, walk 10 feet, turn around and sit back down in the same chair.

SECONDARY OUTCOMES:
Falls Self-Efficacy | Baseline to 16 weeks
  The confidence a person has in their ability to walk without falling measured via a 10-item Likert -type 10-point scale with score ranges from 10-100, where 10 is low confidence and 100 is high confidence in their ability to perform various activities without falling.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah L Szanton, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Szanton SL, Clemson L, Liu M, Gitlin LN, Hladek MD, LaFave SE, Roth DL, Marx KA, Felix C, Okoye SM, Zhang X, Bautista S, Granbom M. Pilot Outcomes of a Multicomponent Fall Risk Program Integrated Into Daily Lives of Community-Dwelling Older Adults. J Appl Gerontol. 2021 Mar;40(3):320-327. doi: 10.1177/0733464820912664. Epub 2020 Mar 20. PMID 32193981
- [Derived] Granbom M, Clemson L, Roberts L, Hladek MD, Okoye SM, Liu M, Felix C, Roth DL, Gitlin LN, Szanton S. Preventing falls among older fallers: study protocol for a two-phase pilot study of the multicomponent LIVE LiFE program. Trials. 2019 Jan 3;20(1):2. doi: 10.1186/s13063-018-3114-5. PMID 30606239